CLINICAL TRIAL: NCT02998788
Title: Risk Evaluation and Management in Heart Failure
Acronym: REM-HF
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Wei Jin, Professor,Department of Cardiology, Ruijin Hospital
Other Study IDs: RJ-81600198
Record Dates: First submitted 2016-12-10; First posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Heart Failure; Risk Factor, Cardiovascular
Keywords: heart failure; risk factor; cardiovascular disease; lifestyle behavior
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fasting (8-12 hours) venous blood samples were drawn and transfused into vacuum tubes containing EDTA during the study visits. These samples were stored and further analyzed in the Central Laboratory of Ruijin Hospital.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is an prospective study conducted in a Chinese heart failure population. The study investigates the effects of cardiovascular disease risk factors such as lifestyle behaviors,biomarkers and intermediate diseases on heart failure prognosis.

DETAILED DESCRIPTION:
Heart failure is the main cause of cardiovascular death. The primary goal of this study is to estimate the association of lifestyle behavior (e.g., alcohol, tea and coffee consumption, sedentary behavior, smoking habit, sleep disorder and physical activity), intermediate conditions (e.g., hypertension, diabetes and dyslipidemia), genetic risk factors and circulating biomarkers with heart failure prognosis. Another goal is to improve the health status and reduce cardiovascular events and death for heart failure patients via patient education, disease monitoring and medication titration. This study planned to consecutively enroll 1,000 heart failure patients fulfilling the inclusion criteria. Each participants will be followed up for at least 5 years. The study endpoints, all-cause mortality and cardiovascular events, will be identified by directly contacting participants during the follow-up surveys, checking pertinent medical records and discharge lists from the hospitals, or checking death certificates from local vital statistics offices. The Cox proportional hazard model will be used to estimate the risk factors for health outcomes in heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 and above
* inpatient with one of the following clinical situations:

  * congestive heart failure (pulmonary edema,pulmonary congestion or peripheral edema)
  * cardiogenic shock
  * Insufficient high output cardiac
* with impaired cardiac function diagnosed by echocardiography
* able to provide informed consent

Exclusion Criteria:

* expressed refusal to participate in the baseline investigation or follow-up visits Severe co-morbidity associated with a reduction in life expectancy of less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with primary discharge diagnosis of heart failure
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-06; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 10 years
A composite of cardiovascular events | 10 years
  A composite of myocardial infarction, revascularization, stroke, rehospitalization due to heart failure and cardiovascular death

SECONDARY OUTCOMES:
myocardial infarction | 10 years
revascularization | 10 years
stroke | 10 years
rehospitalization due to heart failure | 10 years
cardiovascular death | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jin, Professor, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided